CLINICAL TRIAL: NCT03584776
Title: A Randomized Controlled Trial of Virtual Reality for Pain Management in the Post-Operative Period Following Orthopedic Surgery
Brief Title: Virtual Reality for Post-operative Pain Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gillette Children's Specialty Healthcare (Other)
Responsible Party: Principal Investigator, Chantel Burkitt, Principal Investigator, Gillette Children's Specialty Healthcare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003725
Record Dates: First submitted 2018-06-11; First posted 2018-07-12 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Spinal Fusion
Keywords: Virtual reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Virtual Reality Post Spinal Fusion (Experimental): Patients randomized to the VR group will have the opportunity to utilize VR during the post operative period, and will also experience VR during research visits each day following surgery.
  Interventions: Device: Virtual Reality
- Standard of Care (No Intervention): Patients randomized to the non-VR condition will experience the usual standard of care following spinal fusion surgery. This will include 15-30 minutes of movie viewing during research visits.

INTERVENTIONS:
Device: Virtual Reality — Participants randomized to the VR condition will experience an an immersive guided relaxation VR experience during research visits in the post-operative period. They will also have the opportunity to choose additional VR games and relaxation experiences during their inpatient stay.
  Arms: Virtual Reality Post Spinal Fusion

SUMMARY:
Use an RCT study design to measure pain experience, medication use, medical side effects, and length of hospital stay with and without availability of VR following spine fusion surgery

DETAILED DESCRIPTION:
The purpose of this study is to prospectively assess the utility of virtual reality (VR) for pain and anxiety management in the post-operative period following major orthopedic surgery. While there is substantial evidence supporting the use of VR during dressing changes for burn victims, there is little known about VR use in post-surgical settings. In the proposed study, patients will be randomized to either receive VR in addition to standard of care or to receive only standard of care during their post-operative care following spinal fusion surgery for idiopathic scoliosis or neuromuscular scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is having a spinal fusion at Gillette Children's Specialty Healthcare
* Patient with a diagnosis of adolescent idiopathic scoliosis (AIS) or a diagnosis of neuromuscular scoliosis

Exclusion Criteria:

* Non-English speaking parents/patients
* Patients with history of motion sickness
* Patients with epilepsy
* Patients with a ventricular shunt
* Patients with severe/profound cognitive impairments

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Timing of pain medication | 4 days
  Timing of morphine equivalent opioids (mg/kg/day) and adjunctive medications (e.g., Tylenol, Diazepam, Propofol, Midazolam, etc.; mg/kg/day).This will be collected retrospectively from the patient medical record following the conclusion of treatment.
Doses of pain medication | 4 days
  Doses of morphine equivalent opioids (mg/kg/day) and adjunctive medications (e.g., Tylenol, Diazepam, Propofol, Midazolam, etc.; mg/kg/day).This will be collected retrospectively from the patient medical record following the conclusion of treatment.

SECONDARY OUTCOMES:
Parents' Postoperative Pain Measure | 4 days
  The Parents' Postoperative Pain Measure (PPPM-SF) is a measure of pain-related behavioral changes. The PPPM-SF is 10 question yes/no scale, covering functional interference (5 items) and pain behaviors (5 items) and asks parents to compare the child's behaviors with their typical behavior. Each score of "yes" is counted as 1-point, yielding a total score of 0-10 (higher scores indicating higher pain intensity). Parents will complete this measure daily until their child is discharged from the hospital.
Faces Pain Scale-Revised | 4 days
  The Faces Pain Scale-Revised (FPS-R) will be used to assess pain intensity in the post-operative period (for 1-6 days, depending on the length of inpatient stay) for the purposes of this study. The FPS-R will be used to assess pain intensity (faces indicating 0-10 pain scale, 0 face indicating no pain, 10 equals very much pain) "right now" and will be completed by the patient and parent (when present) at the beginning of each daily research visit for both the VR and non-VR groups. The VR group will complete the FPS-R again following the research facilitated VR session. For consistency purposes, parents will also be asked to report their perception of the patient's pain using the FPS-R.
Visual analogue scale | 4 days
  A visual analogue scale (VAS) will be used to quantify multiple aspects of the treatment experience expected to be impacted by the use of VR. The VAS will be a 10 cm 0-100 scale (0 indicating no pain, 100 indicating very much pain), will be completed once per day by both the VR and non-VR groups, and will reflect the past 24 hour period. Participants and their parents in the VR condition will complete the VAS a second time each day following the research facilitated VR experience (second VAS will reflect the past 15 minutes). The VAS will assess the following: patient anxiety; parent anxiety; patient and parent time spent thinking about pain; pain unpleasantness; average pain rating; pain rating right now; worst pain rating; least pain rating; engagement during VR (VR group only); and satisfaction with pain management.
Length of stay | 4 days
  Length of inpatient stay following surgery (collected from medical record)
Pain assessment scores | 4 days
  Nursing pain assessment scores (collected from medical record)
Time patient out of bed | 4 days
  Duration of time from surgery to patient out of bed and walking (collected from medical record).

CONTACTS AND LOCATIONS:
Overall Officials: Chantel Barney, PhD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li L, Yu F, Shi D, Shi J, Tian Z, Yang J, Wang X, Jiang Q. Application of virtual reality technology in clinical medicine. Am J Transl Res. 2017 Sep 15;9(9):3867-3880. eCollection 2017. PMID 28979666
- [Background] Hoffman HG, Doctor JN, Patterson DR, Carrougher GJ, Furness TA 3rd. Virtual reality as an adjunctive pain control during burn wound care in adolescent patients. Pain. 2000 Mar;85(1-2):305-9. doi: 10.1016/s0304-3959(99)00275-4. PMID 10692634
- [Background] Schmitt YS, Hoffman HG, Blough DK, Patterson DR, Jensen MP, Soltani M, Carrougher GJ, Nakamura D, Sharar SR. A randomized, controlled trial of immersive virtual reality analgesia, during physical therapy for pediatric burns. Burns. 2011 Feb;37(1):61-8. doi: 10.1016/j.burns.2010.07.007. Epub 2010 Aug 7. PMID 20692769
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Asl Aminabadi N, Erfanparast L, Sohrabi A, Ghertasi Oskouei S, Naghili A. The Impact of Virtual Reality Distraction on Pain and Anxiety during Dental Treatment in 4-6 Year-Old Children: a Randomized Controlled Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2012 Fall;6(4):117-24. doi: 10.5681/joddd.2012.025. Epub 2012 Nov 12. PMID 23277857
- [Background] Hua Y, Qiu R, Yao WY, Zhang Q, Chen XL. The Effect of Virtual Reality Distraction on Pain Relief During Dressing Changes in Children with Chronic Wounds on Lower Limbs. Pain Manag Nurs. 2015 Oct;16(5):685-91. doi: 10.1016/j.pmn.2015.03.001. Epub 2015 May 9. PMID 25972074
- [Background] Jones T, Moore T, Choo J. The Impact of Virtual Reality on Chronic Pain. PLoS One. 2016 Dec 20;11(12):e0167523. doi: 10.1371/journal.pone.0167523. eCollection 2016. PMID 27997539
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Background] Steele E, Grimmer K, Thomas B, Mulley B, Fulton I, Hoffman H. Virtual reality as a pediatric pain modulation technique: a case study. Cyberpsychol Behav. 2003 Dec;6(6):633-8. doi: 10.1089/109493103322725405. PMID 14756928
- [Background] Cacau Lde A, Oliveira GU, Maynard LG, Araujo Filho AA, Silva WM Jr, Cerqueria Neto ML, Antoniolli AR, Santana-Filho VJ. The use of the virtual reality as intervention tool in the postoperative of cardiac surgery. Rev Bras Cir Cardiovasc. 2013 Jun;28(2):281-9. doi: 10.5935/1678-9741.20130039. PMID 23939326
- [Background] Bieri D, Reeve RA, Champion DG, Addicoat L, Ziegler JB. The Faces Pain Scale for the self-assessment of the severity of pain experienced by children: development, initial validation, and preliminary investigation for ratio scale properties. Pain. 1990 May;41(2):139-150. doi: 10.1016/0304-3959(90)90018-9. PMID 2367140
- [Background] Ramstad K, Jahnsen R, Skjeldal OH, Diseth TH. Characteristics of recurrent musculoskeletal pain in children with cerebral palsy aged 8 to 18 years. Dev Med Child Neurol. 2011 Nov;53(11):1013-8. doi: 10.1111/j.1469-8749.2011.04070.x. PMID 22014321
- [Background] Hoffman HG, Patterson DR, Carrougher GJ. Use of virtual reality for adjunctive treatment of adult burn pain during physical therapy: a controlled study. Clin J Pain. 2000 Sep;16(3):244-50. doi: 10.1097/00002508-200009000-00010. PMID 11014398
- [Background] Sharar SR, Miller W, Teeley A, Soltani M, Hoffman HG, Jensen MP, Patterson DR. Applications of virtual reality for pain management in burn-injured patients. Expert Rev Neurother. 2008 Nov;8(11):1667-74. doi: 10.1586/14737175.8.11.1667. PMID 18986237
- [Background] Hoffman HG, Seibel EJ, Richards TL, Furness TA, Patterson DR, Sharar SR. Virtual reality helmet display quality influences the magnitude of virtual reality analgesia. J Pain. 2006 Nov;7(11):843-50. doi: 10.1016/j.jpain.2006.04.006. PMID 17074626
- [Background] Hoffman HG, Sharar SR, Coda B, Everett JJ, Ciol M, Richards T, Patterson DR. Manipulating presence influences the magnitude of virtual reality analgesia. Pain. 2004 Sep;111(1-2):162-8. doi: 10.1016/j.pain.2004.06.013. PMID 15327820
- [Background] von Baeyer CL, Chambers CT, Eakins DM. Development of a 10-item short form of the parents' postoperative pain measure: the PPPM-SF. J Pain. 2011 Mar;12(3):401-6. doi: 10.1016/j.jpain.2010.10.002. Epub 2010 Dec 17. PMID 21167790
- [Background] Chambers CT, Finley AG, McGrath PJ, Walsh TM. The parents' postoperative pain measure: replication and extension to 2-6-year-old children. Pain. 2003 Oct;105(3):437-443. doi: 10.1016/S0304-3959(03)00256-2. PMID 14527704
- [Background] Hoffman HG, Richards TL, Coda B, Bills AR, Blough D, Richards AL, Sharar SR. Modulation of thermal pain-related brain activity with virtual reality: evidence from fMRI. Neuroreport. 2004 Jun 7;15(8):1245-8. doi: 10.1097/01.wnr.0000127826.73576.91. PMID 15167542
- [Background] Wittwer A, Krummenacher P, La Marca R, Ehlert U, Folkers G. Salivary Alpha-Amylase Correlates with Subjective Heat Pain Perception. Pain Med. 2016 Jun;17(6):1131-6. doi: 10.1093/pm/pnv085. Epub 2016 Jan 13. PMID 26764337
- [Background] Shinde SK, Danov S, Chen CC, Clary J, Harper V, Bodfish JW, Symons FJ. Convergent validity evidence for the Pain and Discomfort Scale (PADS) for pain assessment among adults with intellectual disability. Clin J Pain. 2014 Jun;30(6):536-43. doi: 10.1097/AJP.0000000000000020. PMID 24135902
- [Background] Phan A, Edwards CL, Robinson EL. The assessment of pain and discomfort in individuals with mental retardation. Res Dev Disabil. 2005 Sep-Oct;26(5):433-9. doi: 10.1016/j.ridd.2004.10.001. PMID 16039095
- [Background] Norton M, Holm JE, McSherry WC 2nd. Behavioral assessment of relaxation: the validity of a Behavioral Rating Scale. J Behav Ther Exp Psychiatry. 1997 Jun;28(2):129-37. doi: 10.1016/s0005-7916(97)00004-9. PMID 9194010
- [Background] Pielech M, Ryan M, Logan D, Kaczynski K, White MT, Simons LE. Pain catastrophizing in children with chronic pain and their parents: proposed clinical reference points and reexamination of the Pain Catastrophizing Scale measure. Pain. 2014 Nov;155(11):2360-7. doi: 10.1016/j.pain.2014.08.035. Epub 2014 Aug 29. PMID 25180013
- [Background] Breau LM, Camfield CS, McGrath PJ, Finley GA. The incidence of pain in children with severe cognitive impairments. Arch Pediatr Adolesc Med. 2003 Dec;157(12):1219-26. doi: 10.1001/archpedi.157.12.1219. PMID 14662579
- [Background] Barney CC, Krach LE, Rivard PF, Belew JL, Symons FJ. Motor function predicts parent-reported musculoskeletal pain in children with cerebral palsy. Pain Res Manag. 2013 Nov-Dec;18(6):323-7. doi: 10.1155/2013/813867. PMID 24308022
- [Background] Engel JM, Kartin D, Carter GT, Jensen MP, Jaffe KM. Pain in youths with neuromuscular disease. Am J Hosp Palliat Care. 2009 Oct-Nov;26(5):405-12. doi: 10.1177/1049909109346165. PMID 19820205
- [Background] Symons FJ, Rivard PF, Nugent AC, Tervo RC. Parent evaluation of spasticity treatment in cerebral palsy using botulinum toxin type A. Arch Phys Med Rehabil. 2006 Dec;87(12):1658-60. doi: 10.1016/j.apmr.2006.08.343. PMID 17141650
- [Background] Fernandez-Blazquez MA, Avila-Villanueva M, Lopez-Pina JA, Zea-Sevilla MA, Frades-Payo B. Psychometric properties of a new short version of the State-Trait Anxiety Inventory (STAI) for the assessment of anxiety in the elderly. Neurologia. 2015 Jul-Aug;30(6):352-8. doi: 10.1016/j.nrl.2013.12.015. Epub 2014 Jan 28. English, Spanish. PMID 24484757
- [Background] Perpina-Galvan J, Richart-Martinez M, Cabanero-Martinez MJ, Martinez-Dura I. Content validity of the short version of the subscale of the State-Trait Anxiety Inventory (STAI). Rev Lat Am Enfermagem. 2011 Jul-Aug;19(4):882-7. doi: 10.1590/s0104-11692011000400005. English, Portuguese, Spanish. PMID 21876939